CLINICAL TRIAL: NCT02050230
Title: Hemodynamic Effects of Stored Blood Transfusion in Intensive Care Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Protracted recruitment of patients
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, David M Baron, MD, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BASG 2013-002316-27; 2013-002316-27 (EudraCT Number)
Record Dates: First submitted 2014-01-17; First posted 2014-01-30 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Hypertension
Keywords: transfusion; pulmonary hypertension; intensive care medicine
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Blood Transfusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fresh blood transfusion (Active Comparator): One unit of blood stored for less than 14 days
  Interventions: Biological: Blood transfusion
- Standard issue blood transfusion (Experimental): One unit of blood stored under standard conditions
  Interventions: Biological: Blood transfusion

INTERVENTIONS:
Biological: Blood transfusion — One unit of red blood cells will be transfused over the course of 20 minutes

SUMMARY:
Transfusion of stored blood has been associated with increased pulmonary vascular resistance in lambs. The investigators hypothesize that transfusion of one unit of red blood cells stored under standard conditions in intensive care patients will increase pulmonary arterial pressure and pulmonary vascular resistance to a greater extent than will one unit of fresh red blood cells.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a pulmonary artery catheter in place
2. Transfusion of 1 unit of packed red blood cells indicated for standard intensive care therapy
3. The patient has an arterial catheter

Exclusion Criteria:

1. Age < 18 years
2. Clinical prediction that the patient will not survive at least 48 hours
3. Acute bleeding: > 2 units of packed red blood cells/hour
4. Vasopressor use: noradrenalin > 0.2 μg/kg/min or any use of adrenalin within 6 hours of inclusion into the study
5. Therapy with inhaled NO, inhaled prostacyclin, or phosphodiesterase-5-inhibitors
6. Sepsis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pulmonary arterial pressure | Change from baseline to immediately after transfusion (time frame of 20 min)
Pulmonary vascular resistance | Change from baseline to immediately after transfusion (time frame of 20 min)

SECONDARY OUTCOMES:
Systemic pressure | Change from baseline to immediately after transfusion (time frame of 20 min)
Systemic vascular resistance | Change from baseline to immediately after transfusion (time frame of 20 min)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ullrich, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- General Hospital of the Medical University of Vienna, Vienna, Austria